CLINICAL TRIAL: NCT01281111
Title: A Randomized, Double-Blind, Placebo-Controlled Study of the Safety, Tolerability, and Pharmacokinetics of BG00012 Administered With and Without 325 mg Aspirin in Healthy Adult Volunteers
Brief Title: Alternate Dosing Regimens of BG00012 in Healthy Volunteers
Acronym: 109HV106
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: 109HV106
Record Dates: First submitted 2011-01-20; First posted 2011-01-21 (Estimated); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Healthy
MeSH Terms: interventions — Dimethyl Fumarate; Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- BG00012 plus ASA (Experimental)
  Interventions: Drug: Dimethyl Fumarate (BG00012); Drug: Aspirin
- BG00012 plus ASA matching placebo (Experimental)
  Interventions: Drug: Dimethyl Fumarate (BG00012); Drug: ASA matching placebo
- BG00012 Placebo plus ASA (Placebo Comparator)
  Interventions: Drug: Aspirin; Drug: BG00012 matching placebo
- BG00012 Placebo plus ASA matching placebo (Experimental)
  Interventions: Drug: BG00012 matching placebo; Drug: ASA matching placebo
- BG00012 (Experimental): modified dose regimen
  Interventions: Drug: Dimethyl Fumarate (BG00012)

INTERVENTIONS:
Drug: Dimethyl Fumarate (BG00012)
  Arms: BG00012; BG00012 plus ASA; BG00012 plus ASA matching placebo
Drug: Aspirin
  Arms: BG00012 Placebo plus ASA; BG00012 plus ASA
Drug: BG00012 matching placebo
  Arms: BG00012 Placebo plus ASA; BG00012 Placebo plus ASA matching placebo
Drug: ASA matching placebo
  Arms: BG00012 Placebo plus ASA matching placebo; BG00012 plus ASA matching placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and PK of different doses and dosing regimens of BG00012 administered with and without ASA compared to placebo

DETAILED DESCRIPTION:
Preclinical safety margins for BG00012 allow for a maximum daily dose of 720 mg daily. The study will use a variety of clinical scales, including a flushing scale derived from a validated questionnaire [Norquist 2007], to better understand the safety and tolerability of several doses and dosing regimens of BG00012 up to a total daily dose of 720 mg. The etiology of BG00012-induced flushing will be assessed by collecting relevant biomarker data and the impact of ASA on flushing will be evaluated. Assessments relating to GI symptoms will also be performed.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information (PHI) in accordance with national and local subject privacy regulations.
* Aged 18 to 55 years old, inclusive, at the time of informed consent.
* Must be in good health, as determined by the Investigator, based on medical history and screening evaluations.
* Must have a body mass index of 18 to 34 kg/m2, inclusive.
* Subjects of childbearing potential must practice effective contraception during the study and be willing and able to continue contraception for 30 days after their last dose of study treatment.

Exclusion Criteria:

* History of any clinically significant cardiac, endocrinologic, GI, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal, or other major disease, as determined by the Investigator.
* History of malignant disease, including solid tumors and hematologic malignancies (except basal cell and squamous cell carcinomas of the skin that have been completely excised and are considered cured).
* Serious infection (e.g., pneumonia, septicemia) as determined by the Investigator within the 3 months prior to Day 1.
* Diarrhea, constipation, abdominal pain, flushing, or nausea within 28 days prior to Day 1.
* History of severe allergic or anaphylactic reactions. Additionally, subjects with a history of intolerance to ASA or non-steroidal anti-inflammatory drugs (NSAIDS) must be excluded.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2011-02-01 (Actual); Primary Completion 2011-03-18 (Actual); Study Completion 2011-03-18 (Actual)

PRIMARY OUTCOMES:
• incidence of treatment emergent AEs | 11 days
• incidence of serious AEs (SAEs) | 11 days
• clinical laboratory assessments: | 11 days
• Concentration versus time data for BG00012 (as measured by monomethyl fumarate (MMF), will be collected for each treatment group. Plasma PK parameters will include AUC, Cmax, time to maximum plasma concentration, half life & lagtime. | 11 days

SECONDARY OUTCOMES:
• incidence, severity, and duration (time of onset until time of resolution) of flushing based on flushing severity measurements. | 11 days
• Incidence, severity, duration, and characteristics of GI events | 11 days
• concentrations of PGD2 and/or its metabolites in plasma and/or urine and other prostaglandins, as well as other biomarkers in plasma and/or urine | 11 days

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Saint Paul, Minnesota, United States

REFERENCES:
- [Derived] Sheikh SI, Nestorov I, Russell H, O'Gorman J, Huang R, Milne GL, Scannevin RH, Novas M, Dawson KT. Tolerability and pharmacokinetics of delayed-release dimethyl fumarate administered with and without aspirin in healthy volunteers. Clin Ther. 2013 Oct;35(10):1582-1594.e9. doi: 10.1016/j.clinthera.2013.08.009. PMID 24139424